CLINICAL TRIAL: NCT01963936
Title: NEWBORN VENTILATION IN THE DELIVERY ROOM: CAN IT BE IMPROVED WITH A LARYNGEAL MASK AIRWAY? A Prospective, Randomized Single-center Study
Brief Title: Supreme-LMA for Neonatal Resuscitation: a Prospective, Randomized Single-center Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Donato Nitti, Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLMA in neonatal resuscitation
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Neonatal Resuscitation
Keywords: Infant newborn; Laryngeal mask airway; Positive pressure ventilation; Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supreme LMA (Experimental)
  Interventions: Device: Supreme LMA
- Facial mask (Active Comparator)
  Interventions: Device: Facial mask

INTERVENTIONS:
Device: Supreme LMA
  Arms: Supreme LMA
Device: Facial mask
  Arms: Facial mask

SUMMARY:
Laryngeal mask airways (LMA) that fit over the laryngeal inlet have been shown to be effective for ventilating newborns at birth. The LMA may be considered as an alternative to FM for positive pressure ventilation (PPV) among newborns weighing >2000 g or delivered >34 weeks' gestation.

A recent, quasi-experimental study provided the feasibility, efficacy and safety of using the LMA in neonatal resuscitation.

However, studies of LMA use for providing PPV during neonatal resuscitation are still limited. There are no published clinical randomized trials evaluating the LMA compared with the FM for neonatal resuscitation.

Hypothesis: Our hypothesis is based on the assumption that ventilating newborns needing PPV with a LMA will be more effective than ventilating with a FM by decreasing the proportion of resuscitated newborns needing ETT.

Objective: To compare the effectiveness of LMA and FM ventilation in newborns needing PPV at birth.

Design / Methods: An open, prospective, randomized, single center, clinical trial.

Intervention: PPV will be performed with a LMA (intervention group) or with a FM (control group) in all infant newborns weighing >2000 g or delivered >34 weeks gestation.

Primary outcome variable: Proportion of newborns needing endotracheal intubation.

Secondary outcome measures: Apgar score at 5 minutes, heart rate at 60, 90 seconds and 5 and 10 minutes, time to first breath, duration of PPV, for proportion of infants needing chest compressions, drugs and death within 1 week and/or presence of HIE, grade II or III, according to a modification of Sarnat and Sarnat.2,10 According to this classification, HIE grade I (mild) includes irritability, hyperalertness, mild hypotonia, and poor sucking; grade II (moderate) includes lethargy, seizures, marked abnormalities of tone, and requirement of tube feeding; and grade III (severe) includes coma, prolonged seizures, severe hypotonia, and failure to maintain spontaneous respiration.

The following data were collected during resuscitation: (1) Apgar score at 1 min and 5 min after birth; (2) LMA insertion time, the rate of successful insertion at the first attempt, and the number of attempts required to insert the LMA successfully; (3) duration of resuscitation: response time (the time period from starting LMA resuscitation to achieving an effective response), ventilation time; (4) adverse effects during resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Infants with gestational age ≥34 weeks, an expected birth weight >1.500 g, needing positive pressure ventilation at birth.

Exclusion Criteria:

* Lethal anomalies, hydrops, major malformations of the respiratory system, congenital heart disease, and stillbirths

Max Age: 5 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of newborns needing endotracheal intubation | 10 minutes of life

SECONDARY OUTCOMES:
Time to first breath | 30 minutes of life
Proportion of patients needing Chest compressions and medications | 30 minutes of life
Proportion of patients with hypoxic ischemic encephalopathy | 1 week of life

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neonatal Intensive Care, Hanoi, Vietnam

REFERENCES:
- [Derived] Trevisanuto D, Cavallin F, Nguyen LN, Nguyen TV, Tran LD, Tran CD, Doglioni N, Micaglio M, Moccia L. Supreme Laryngeal Mask Airway versus Face Mask during Neonatal Resuscitation: A Randomized Controlled Trial. J Pediatr. 2015 Aug;167(2):286-91.e1. doi: 10.1016/j.jpeds.2015.04.051. Epub 2015 May 21. PMID 26003882
- [Derived] Trevisanuto D, Cavallin F, Mardegan V, Loi NN, Tien NV, Linh TD, Chien TD, Doglioni N, Chiandetti L, Moccia L. LMA Supreme for neonatal resuscitation: study protocol for a randomized controlled trial. Trials. 2014 Jul 15;15:285. doi: 10.1186/1745-6215-15-285. PMID 25027230